CLINICAL TRIAL: NCT04405687
Title: Post-reconstructive Surgeries of Severe Head and Face Deformities: An Observational Follow-up Study
Brief Title: Postoperative Follow up After Head and Face Reconstructive Surgeries
Status: Completed | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, zantao, Researcher of Plastic and Reconstructive Surgery, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: Follow Up
Record Dates: First submitted 2020-05-25; First posted 2020-05-28 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Deformity of Face

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe head and face deformity
  Interventions: Procedure: Severe head and face deformity reconstructive surgery

INTERVENTIONS:
Procedure: Severe head and face deformity reconstructive surgery — Three questionnaires, including the 36-Item Short Form Health Survey questionnaire (SF-36), Aesthetic and Functional Status Score of Facial Soft-Tissue Deformities/Defects (A&F) and Euroqol 5 dimensions 5 levels questionnaire (EQ-5D-5L), were conducted to evaluate their quality of life and satisfaction with facial aesthetic and functional status.

SUMMARY:
In this observational follow-up study, patients with type III-IV head and face soft tissue deformities/defects following reconstructive surgeries will be asked to fill out 3 questionnaires, either through phone calls or video calls, in order to evaluate the post-operative outcomes such as morphological and functional recovery, quality of life and patients' return to the community.

DETAILED DESCRIPTION:
The objective of this follow up study is to evaluate the effectiveness and to analyze the limitations of the existing management and treatment of severe burn injuries. Investigation of the factors affecting the recovery and patients' return to the community in patients with severe burn injury may lead to effective amendments of the existing management, and thus aiding in the development of an integrated diagnosis and treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative facial soft tissue deformities/defects of type III and IV
2. Major reconstructive surgery of the head and neck (flap transfer with revision at least once) performed before January 1, 2019.
3. Agreed and able to cooperate with the follow-ups, with signed informed consent form or audio recorded informed consent.

Exclusion Criteria:

1. Patients with mental illness, reduced cognitive capacity, unable to consent and unable to cooperate.
2. Minor patients without legal guardian.
3. Not willing to participate; informed consent form not signed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This clinical study will include patients treated by Prof. Li Qingfeng 's professional team who have undergone major head and face reconstructive surgeries before January 1, 2019.
  It is estimated that about 85 patients will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-04-18 (Actual); Study Completion 2020-04-18 (Actual)

PRIMARY OUTCOMES:
SF-36 total score | 12 minutes
  8 aspects including actual physiological function, desirable physiological function, somatic pain, general health status, vitality, social function, emotional function, mental health; and 1 health indicator(reported health transition) Score ranges from 1-100 for each aspects, with higher score indicating a better quality of life.
Aesthetic & Functional total score (Patient edition) | 8 minutes
  3 marks for each aspect; Score ranges from 0-18 for aesthetic status, and 0-21 for functional status, with higher score indicating a better outcome.
  For overall satisfaction of aesthetic and functional status preoperatively and postoperatively, score ranges from 0-10, with higher score indicating a better outcome.
EQ-5D-5L total score | 2 minutes
  Assessment of the patients' mobility, self-care, usual activities, pain/discomfort, anxiety/depression.
  Score ranges from 0-100, with higher score indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zan, MD, PhD, Study Director — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided